CLINICAL TRIAL: NCT04446780
Title: Mediolateral Episiotomy and Prevention of Obstetric Anal Sphincter Injuries in Instrumental Delivery: a Prospective Population-based Propensity Score Study
Brief Title: Mediolateral Episiotomy and Obstetric Anal Sphincter Injuries in Instrumental Delivery
Acronym: INSTRUMODA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: INSTRUMODA
Record Dates: First submitted 2020-06-15; First posted 2020-06-25 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-04

CONDITIONS: Obstetric Anal Sphincter Injury; Episiotomy Wound; Anal Incontinence; Pelvic Floor Disorders; Depression
MeSH Terms: conditions — Encopresis; Pelvic Floor Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women who underwent an episiotomy: Nulliparous women who underwent an instrumental vaginal delivery with mediolateral episiotomy
  Interventions: Procedure: Mediolateral episiotomy
- Women who did not underwent an episiotomy: Nulliparous women who underwent an instrumental vaginal delivery without mediolateral episiotomy

INTERVENTIONS:
Procedure: Mediolateral episiotomy — Cutting of the perineum during vaginal delivery in order to avoid obstetric anal sphincter injury
  Groups: Women who underwent an episiotomy

SUMMARY:
Literature is contradictory about the impact of mediolateral episiotomy during operative vaginal delivery in obstetric anal sphincter injuries prevention explaining the absence of international guidelines. The investigators consider that a randomized trials does not appears feasible for both ethical and practical reason and so we suggest a large national observational study.

The investigators will include all nulliparous women that underwent an operative vaginal delivery within the 72h following the delivery at more than 34 weeks of amenorrhea. The investigators will collect data about the history of pregnancy, the course of labor, the mode of delivery, maternal immediate and one-year morbidity, neonatal immediate morbidity. The investigators expect a one-year study in 129 recruiting center with 15000 included women.

The primary objective is to assess the protective effect of mediolateral episiotomy against obstetric anal sphincter injury during instrumental delivery in nulliparous women according to the type of instrument used. The secondary endpoints are to investigate the effect of mediolateral episiotomy on one-year maternal morbidity, immediate maternal morbidity. The investigators also aim to develop a clinical score to assess the absolute risk of obstetric anal sphincter injury during instrumental delivery. Finally, the investigators will investigate the impact of fetal presentation ultrasound assessment immediately before instrumental delivery on the mode of delivery.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 years or older
* nulliparity and instrumental delivery of a singleton in cephalic presentation in the previous 72 hours including failure of vaginal instrumental delivery leading to cesarean section

Exclusion Criteria:

* expression of any opposition or objection to study participation
* previous delivery of a fetus at a gestational age greater than 20 weeks, regardless of the mode of delivery
* preterm birth before 34 weeks of amenorrhea
* fetal presentation other than cephalic
* multiple pregnancy
* in utero death
* inability to understand French
* under judicial protection
* without access to a numeric terminal with internet connexion

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will include in 121 centers in France during women year women who gave birth to their first child with requirement of an operative delivery. We will compare those who underwent a mediolateral episiotomy to those wo have not for the occurrence of obstetric anal sphincter injury according to the type of instrument used
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Obstetric Anal Sphincter Injury (mediolateral episiotomy vs no episiotomy for each type of instrument) | Immediately after the delivery
  Perineal tears involving the anal sphincter complex (3rd and 4th degree according RCOG OMS classification)

SECONDARY OUTCOMES:
Immediate maternal morbidity (mediolateral episiotomy vs no episiotomy) | through mother's hospitalization, an average of 4 days
  post partum hemorrhage, perineal infection, perineal hematoma, perineal pain, difficulty for voiding, satisfaction about childbirth, intensive care admission, death
Immediate neonatal morbidity (mediolateral episiotomy versus no episiotomy) | through mother's hospitalization, an average of 4 days
  Clinical vitality status, neonatal cephalic marks , neonatal bone fractures, admission into intensive unit care, death
One year maternal morbidity (mediolateral episiotomy versus no episiotomy) | 1 year
  Anal incontinence, urinary incontinence, perineal pain, postnatal depression, sexual function, self rated health
Association between fetal presentation assessment before the delivery and the issue of delivery (ultrasound assessment versus no ultrasound assessment) | through mother's hospitalization, an average of 4 days
  Failed instrumental delivery defined as a requirement of several instrument and/or requirement of cesarean section
Development of a clinical score to assess the absolute risk of obstetric anal sphincter injury during instrumental delivery (with or without mediolateral episiotomy) | through mother's hospitalization, an average of 4 days
  We will report the sensitivity, specificity and area under the curve of this score.

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital, Poitiers, France

REFERENCES:
- [Derived] Gachon B, Durocher L, Garabedian C, Guerby P, Chauleur C, Bertholdt C, Desplanches T, Sentilhes L, Sibiude J, Mottet N, Le Ray C, Estzo ML, Lassel L, Bel S, Devouge P, Dochez V, Riethmuller D, Schmitz T, Vincent-Rohfritsch A, Harvey T, Delaunay F, Ducarme G, Checchi-Guichard C, Foucher Y, de Tayrac R, Pizzoferrato AC, Pierre F, Berveiller P, Fritel X; INSTRUMODA Study Group; GROG (Groupe de Recherche en Obstetrique et Gynecologie). Episiotomy to prevent obstetric anal sphincter injuries during instrumental delivery in nulliparous women: a national prospective comparative cohort study. Am J Obstet Gynecol. 2025 Aug;233(2):123.e1-123.e24. doi: 10.1016/j.ajog.2025.01.029. Epub 2025 Jan 30. PMID 39889841
- [Derived] Gachon B, Schmitz T, Artzner F, Parant O, De Tayrac R, Ducarme G, Le Ray C, Pizzoferrato AC, Garabedian C, Riethmuller D, Pierre F, Ragot S, Fritel X; GROG (Groupe de Recherche en Gynecologie Obstetrique). A core outcome set development for a French national prospective study about the effect of mediolateral episiotomy on obstetric anal sphincter injury during operative vaginal delivery (INSTRUMODA). BMC Pregnancy Childbirth. 2021 Mar 25;21(1):251. doi: 10.1186/s12884-021-03603-0. PMID 33765964